CLINICAL TRIAL: NCT02742337
Title: Identification of Epigenetic Biomarkers for Early Detection of Rheumatic Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arthritis Northwest PLLC (Industry)
Collaborators: Epigenesys LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: AE010831
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Epigenetic
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Specimens Collected:
  1. Blood: Monocytes
  2. Mucosal Swab: Buccal cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test: Newly diagnosed female patients with rheumatoid arthritis who have not previously used a disease modifying anti-rheumatic drug.
- Control: Female patients not having a diagnosis of rheumatoid arthritis and who have not previously used a disease modifying anti-rheumatic drug.

SUMMARY:
• Given the cost and risk associated with biologic disease modifying anti-rheumatic drugs (bDMARDs), selection of the optimal medication is imperative. Current attempts to identify genetic factors that predict bDMARD response and effectiveness in rheumatoid arthritis patients have been inconclusive. Furthermore the presence of epigenetic signatures in rheumatoid arthritis patients has not been established. This protocol is the first step to identifying the practicality and feasibility of epigenetic testing to aid in diagnosis and/or medication selection in rheumatoid arthritis patients. Subsequent research into such epigenetic changes may be indicative of bDMARD response and/or safety. If such epigenetic signatures (EGS) exist the business need for such tests will thus be supported.

DETAILED DESCRIPTION:
Two groups of patients will be assessed for the presence unique epigenetic signatures. The test group, having a bonafide diagnosis of rheumatoid arthritis (RA) and a control group of subjects who does not fulfill the American College of Rheumatology's classification criteria for RA. A buccal cell sample and blood draw will be sequenced and analyzed from each subject in each group for the presence of epigenetic signatures.

ELIGIBILITY:
Test patient Inclusion Criteria:

* Must fulfill the 2010 ACR rheumatoid arthritis classification criteria.
* Must have at least moderate disease activity (CDAI) for most recent disease activity score
* Any history of NSAID or corticosteroid use is acceptable
* Weight at time of blood draw must be greater than 110 lbs.
* Must be RF+ or CCP+

Control patient Inclusion Criteria:

* Female (age: 18 - 80)
* Must not fulfill the 2010 ACR rheumatoid arthritis classification criteria.
* Weight at time of blood draw must be greater than 110 lbs.
* Age will be within 5 years of a test patient.

Exclusion Criteria:

* Male
* Age 17 or less
* History of Disease Modifying Anti-Rheumatic Drugs (DMARDs), or biologic DMARDs.
* History of malignancy, except non-melanoma skin cancer
* Previous treatment for malignancy with chemotherapy agents
* Patient reported history of HIV, HepB, HepC, or TB

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is at-risk patients for chronic auto-immune and rheumatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Counts of patients with epigenetic signatures. | 1 day
  The identification of a statistically significant number of RA patients having a consistent epigenetic signature

CONTACTS AND LOCATIONS:
Locations (1):
- Arthritis Northwest, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No